CLINICAL TRIAL: NCT00383643
Title: Xyrem(Sodium Oxybate) and Ambien(Zolpidem Tartrate) in the Treatment of Chronic Insomnia: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group Study.
Brief Title: Xyrem(Sodium Oxybate) and Ambien(Zolpidem Tartrate) in the Treatment of Chronic Insomnia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jed E Black, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 95900
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem; Sodium Oxybate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Eligible subjects randomized to this arm received placebo as gelatin capsule and a liquid capsule to fully maintain the blind.
  Interventions: Drug: Matching Placebos
- Zolpidem tartrate (Active Comparator): Eligible subjects randomized to this arm received zolpidem as gelatin capsule and a placebo liquid capsule to fully maintain the blind.
  Interventions: Drug: zolpidem tartrate; Drug: Matching Placebos
- Sodium oxybate (Active Comparator): Eligible subjects randomized to this arm received placebo as gelatin capsule and a sodium oxybate capsule to fully maintain the blind.
  Interventions: Drug: sodium oxybate; Drug: Matching Placebos

INTERVENTIONS:
Drug: zolpidem tartrate
  Other Names: Ambien; Zolpidem
  Arms: Zolpidem tartrate
Drug: sodium oxybate
  Other Names: Xyrem
  Arms: Sodium oxybate
Drug: Matching Placebos
  Other Names: Placebo; Sugar pill

SUMMARY:
The primary purpose of the study is to evaluate the long term efficacy of sodium oxybate (Xyrem®) and zolpidem tartrate (Ambien®) in treating chronic insomnia. We will compare the efficacy of sodium oxybate with zolpidem tartrate (Ambien®), and compare the efficacy of each of these two medications with placebos.

DETAILED DESCRIPTION:
Primary aim:

1. To assess the long term efficacy of sodium oxybate and zolpidem tartrate in reducing insomnia and improving sleep quality as assessed by a range of self-reported measures.

Questionnaires and Rating Scales: Subjects completed the following questionnaires and scales: Insomnia Severity Index, Epworth Sleepiness Scale (ESS), Beck Depression Inventory, Pittsburgh Sleep Quality Index (PSQI), Profile of Mood States-Fatigue (POMS). These questionnaires were administered at study baseline, treatment week 4, 8 and 12.

Clinical Global Impression (CGI). The CGI is a clinician-rated scale composed of two subscales that measure disease severity and degree of change, respectively. CGI-Severity (CGI-S) is a single-item, global scale of disease severity that requires the investigator to compare the patient's symptoms with those of all other patients who have the disorder. It is scored from 1 (normal) to 6 (among the most extremely ill of patients). CGI-Change (CGI-C) is a single-item scale of symptomatic improvement or worsening that requires the investigator to compare the patient's status at the time of assessment with baseline severity (baseline CGI-S). One study investigator performed all CGI-S and CGI-C ratings for all subjects.

Randomization. After completing all baseline procedures, eligible subjects were randomized to receive either a combination of active SXB and placebo ZOL (pZOL), active ZOL and placebo SXB (pSXB), or pSXB and pZOL, in a 1:1:1 parallel double-dummy design. A member of the study team who had no contact with subjects and no other role in this study was responsible for preparing study medications according to a randomization schedule. ZOL was encapsulated in lactose powder filled gelatin capsules to be indistinguishable from placebo capsules. Liquid pSXB was designed to match active SXB in appearance, taste and consistency. Subjects were given both liquid and capsule study medications, to maintain the double dummy design. Due to the flexible dose design of this study, subjects and investigators were not blinded to the dosages of study medication/placebo. All subjects were instructed to start study medication at 2.25 grams of SXB/pSXB and 5mg of ZOL/pZOL at bedtime. One study investigator reviewed all potential known side effects of SXB and ZOL prior to dosing, and subjects were instructed to take study medications at the bedside immediately before attempting to sleep, as is the standard administration for SXB.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is obtained.
2. The patient is an outpatient, man or woman of any ethnic origin, 18-75 years of age (inclusive).
3. Patient reports insomnia for at least six months, and insomnia causes the patient distress.
4. The Investigator determines that the patient meets diagnostic criteria for Chronic Insomnia according to International Classification of Sleep Disorders (ICSD) criteria.
5. Sleep diary based screening shows sleep onset latency >30 minutes, and /or wake after sleep onset >30 minutes per night at least 3 nights per week, with combined wake-time-in-bed _> 45 minutes.
6. The patient is in good health as determined by a medical and psychiatric history, and physical examination.
7. Women must be surgically sterile, 2 years post-menopausal, or if of child-bearing potential, using a medically accepted method of birth control, and agree to continued use of this method for the duration of the study.
8. The patient is willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.

Exclusion Criteria:

1. Has any clinically significant, uncontrolled medical or psychiatric conditions. (treated or untreated)
2. Has a probable diagnosis of a current sleep disorder other than Chronic Insomnia.
3. Used any prescription drugs disallowed by the protocol or clinically significant use of over-the counter(OTC) drugs within 14 days before the screening visit.
4. Has a history of alcohol, narcotic, or any other abuse as defined by the DSM-V.
5. Has a clinically significant deviation from normal in the physical examination.
6. Is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)
7. Has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery and succinic semialdehyde dehydrogenase deficiency)
8. Has a known clinically significant drug sensitivity to sodium oxybate or sedative hypnotics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Black, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through local newspaper ads and from the Stanford Sleep Disorders Clinic. A general description of the study was provided. Preliminary screening was conducted by telephone. Interested and qualified persons were scheduled for an in-person screening visit.
Groups:
- Zolpidem Tartrate: Eligible subjects randomized to this arm received zolpidem as a gelatin capsule and a placebo liquid capsule to fully maintain the blind.
- Placebo: Eligible subjects randomized to this arm received placebo (also known as a sugar pill) as gelatin capsule and a liquid capsule to fully maintain the blind.
- Sodium Oxybate: Eligible subjects randomized to this arm received placebo as a gelatin capsule and a sodium oxybate capsule to fully maintain the blind.
Period: Overall Study
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate
Started | 18 | 16 | 14
Completed | 17 | 15 | 13
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate | Total
Number analyzed (Participants) | 18 | 16 | 14 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (9.6) | 56.4 (10.4) | 49.6 (16.3) | 53.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 9 | 32
  Male | 6 | 5 | 5 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Ethnic Minorities | 3 | 5 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 14 | 48

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Clinical Global Impression-change.
Description: Clinician assessment of Clinical Global Impression-Change score at week 12 of treatment intervention. The Clinical Global Impression - Change scale is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the current time point. It is rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. One one clinician provided the ratings in this trial.
Time Frame: Baseline to week 12
Population: All analysis are intent to treat. In the case of missing data, an average value of the available data points (weeks 4 & 8) were used to replace the missing value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate
Number analyzed (Participants) | 18 | 16 | 14
units on a scale | 3.0 (1.2) | 4.2 (1.4) | 2.7 (0.6)

2. Primary Outcome: Assessment of Insomnia Severity Index
Description: Current self-report on Insomnia Severity Index at week 12 of treatment intervention. This is a seven-item questionnaire where the sum of the answers indicate the severity of insomnia. Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate
Number analyzed (Participants) | 18 | 16 | 14
units on a scale | 10.5 (3.9) | 10.8 (6.5) | 8.4 (4.3)

3. Primary Outcome: Assessment of Pittsburgh Sleep Quality Index (PSQI)
Description: Current self-report on Pittsburgh Sleep Quality Index (PSQI) at week 12 of intervention. Consisting of 19 items, the PSQI measures several different aspects of sleep which can be combined into one global score.
  Each item measure is scored on a scale of 0 to 3 where 3 is the extreme negative. The composite PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Based on this questionnaire, a composite score of 5 or greater is indicative of poor sleep quality.
Time Frame: One month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate
Number analyzed (Participants) | 18 | 16 | 14
units on a scale | 8.3 (2.6) | 10.2 (3.5) | 7.9 (2.9)

4. Primary Outcome: Assessment of Fatigue
Description: Current self-report on Profile of Mood State -- Fatigue (POMS-F) at week 12 of intervention. This subscale of the POMS consists of 7 items each scored on a scale of 0 (not at all) to 4 (extremely) which are summed to provide a composite score of fatigue. The range is 0 to 28 for this subscale. Higher scores indicate more fatigue.
Time Frame: One month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate
Number analyzed (Participants) | 18 | 16 | 14
units on a scale | 9.7 (5.4) | 8.0 (7.1) | 5.1 (4.4)

5. Primary Outcome: Assessment of Sleepiness
Description: Current self-report on Epworth Sleepiness Scale (ESS) at week 12 of intervention. This measure consists of 8 scenarios in which the participant is asked to assess how likely s/he is to fall asleep. Scale: 0 = would never doze; 1 = slight chance of dozing; 2 = moderate chance of dozing; 3 = high chance of dozing. Responses are summed for a total score ranging from 0 to 24. The higher the score, the greater the self-reported sleepiness. Scores of 9 and below are considered in the normal range.
Time Frame: One month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate
Number analyzed (Participants) | 18 | 16 | 14
units on a scale | 5.7 (3.7) | 2.9 (2.7) | 4.4 (3.6)

ADVERSE EVENTS:
Arm/Group | Zolpidem Tartrate | Placebo | Sodium Oxybate
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 16/18 | 12/16 | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem Tartrate (N=18) | Placebo (N=16) | Sodium Oxybate (N=15)
seasonal allergy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 2 (2) | 0 (0)
Dry eyes (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Memory (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Pressured speech (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Slow/disorganized speech (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Racing thoughts (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Difficulty with spelling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Coordination/balance (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2)
Disorientation/confusion upon waking (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 10 (10)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Drugged/intoxication feeling (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4)
Groggy/hangover (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Residual/daytime drowsiness (Nervous system disorders) | 9 (9) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 2 (2) | 4 (4)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tinglingness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cramp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Loose stools (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gagging (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 9 (9)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4)
Aches & pains (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 1 (1)
Nocturnia (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Cold (Infections and infestations) | 4 (4) | 4 (4) | 1 (1)
Influenza-like symptom (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gum inflammation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appetite loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Twitch (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmares (General disorders) | 1 (1) | 0 (0) | 1 (1)
Periodic limb movements (General disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep paralysis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional arousal (General disorders) | 0 (0) | 0 (0) | 1 (1)
Snoring (General disorders) | 0 (0) | 0 (0) | 2 (2)
Eating during sleep (General disorders) | 0 (0) | 0 (0) | 1 (1)
Enuresis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bitter aftertaste (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sprained ankle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Insufficient power for most parameters was a planned limitation of the study. Replication with a larger sample is needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No